CLINICAL TRIAL: NCT05861492
Title: The Fatigue Differential Diagnosis Aid (FDDA) for General Practitioners: Utilization Study
Brief Title: FDDA Utilization Study (FDDAU)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment goals could not be met even after amendments to improve recruitment and vast extension of the recruitment period.
Sponsor: Vifor Pharma, Inc. (Industry)
Responsible Party: Sponsor
Organization: Vifor Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: VP-NIS-CH-FFDA-U-05.2016
Record Dates: First submitted 2023-04-11; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-04

CONDITIONS: Fatigue
Keywords: Fatigue; General Practitioner; Differential Diagnosis Aid; PGIC; FDDA; GP
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: Phase 1: Data on current practice was collected by GPs, each providing one patient with unexplained fatigue. None of the GPs used the FDDA.
  Phase 2: The GPs of phase 1 were randomized to two groups (1:1) with half of the GPs in each group.
  Group 1 including additional patients without using the FDDA (control group). Group 2 including additional patients while using the FDDA (experimental group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FDDA Group (Active Comparator): Fatigue anamnesis was done with the help of the Fatigue Differential Diagnosis Aid.
  Interventions: Other: Fatigue Differential Diagnosis Aid
- Non-FDDA group (No Intervention): Fatigue anamnesis was done without the help of the Fatigue Differential Diagnosis Aid.

INTERVENTIONS:
Other: Fatigue Differential Diagnosis Aid — The Fatigue Differential Diagnosis Aid is a systematic questionnaire covering the symptoms and signs of fatigue and the collateral clinical data trying to facilitate the diagnostic process in the care of patient with symptoms of fatigue.
  Arms: FDDA Group

SUMMARY:
This utilization study originally aimed to investigate whether the FDDA could facilitate the differential diagnosis of fatigue and its associated symptoms and consecutively could improve the management and symptoms of fatigue. Furthermore, it aimed at investigating the time until diagnosis, the cause of fatigue, the treatment of fatigue, improvement of fatigue symptoms after treatment, the level of satisfaction of the patients resulting from treatment, time until improvement, improvement of subjective general wellbeing, referrals to other medical specialties and number of visits at physician's office because of fatigue.

The planned endpoints, comparing outcomes in patients diagnosed with and without the help of the FDDA were as follows:

Primary endpoint:

Patient global impression of change (PGIC) at 3 months.

Secondary endpoints:

Patient global impression of change (PGIC) at 6 months; Percentage of patients having experienced a fatigue reduction ≥1 point (NRS); 3 or 6 months after the first visit; Time until an improvement of fatigue ≥1 point (NRS); Mean number of points of fatigue reduction (NRS); Percentage of patients with a PGIC indicating response (=any improvement) after 3 months, 6 months and 3 or 6 months; GP confidence in the established diagnosis; Clinical global impression of change (CGIC); Patient satisfaction of quality of care (diagnosis and treatment); Number of required visits for the same condition; Number of imaging or health services (specialist referrals); required for the diagnosis (MRI, radiograph, etc.); Time to final diagnosis.

DETAILED DESCRIPTION:
Fatigue is a frequently encountered problem in medical practice. It becomes clinically relevant when it is out of proportion, i.e., when it is not obviously caused by objective factors (e.g., excessive workload), but rather occurs as an independent subjective phenomenon manifest in the patient her-/himself, rendering the patient less able to perform daily activities or enjoy recreation adequately.

The Sponsor decided to support an effort to facilitate the diagnostic process in the care of patients with symptoms of fatigue. This implied the creation of a decision aid in the form of a questionnaire covering the symptoms and signs of fatigue and the collateral clinical data (Fatigue Differential Diagnosis Aid, FDDA). The project consists of two studies -the Feasibility Study and the Utilization Study. The Feasibility Study preceded the Utilization Study in order to assess the acceptance and handling properties of the instrument that is used in the Utilization Study.

This study aimed to evaluate the effects of the novel Fatigue Differential Diagnostic Aid (FDDA) in clinical practice and its impact on management of fatigue.

Furthermore, it aimed at investigating the time until diagnosis, the cause of fatigue, the treatment of fatigue, improvement of fatigue symptoms after treatment, the level of satisfaction of the patients resulting from treatment, time until improvement, improvement of subjective general wellbeing, referrals to other medical specialties and number of visits at physician's office because of fatigue.

Study Design:

Prospective, randomized, controlled, multicentre with neither treatment intervention nor study drug.

It was conducted in 2 phases:

Phase 1: Data on current practice was collected by GPs, each providing one patient with unexplained fatigue. None of the GPs used the FDDA. These data were planned to characterize the current practice of diagnosis and treatment choice in patients with unexplained fatigue in the whole study population, to compare patients between both groups of GPs before randomization and to establish the factors used for matching the GP in analysis of primary endpoint in phase 2. Together with data from phase 2 the data were planned to be used for intra-group comparisons.

Phase 2: The GPs of phase 1 were randomized to two groups (1:1) with half of the GPs in each group (inter-group comparison):

Group 1 including additional patients without using the FDDA (control group).

Group 2 including additional patients while using the FDDA (experimental group).

Data concerning patient outcome and number of interventions, quality of care and clinical improvement were collected from the patients and from the treating GPs; data collection time points were at V1 (day 0), V2 (month 1), V3 (month 2), V4 (month 3) and V5 (Month 6); data collection was performed via electronic, or paper based CRF.

The steering committee of the study was composed of experts in the field of fatigue (haematologist, psychosomatician, psychiatrists, epidemiologists, geriatrician, internists, and GP).

The study included patients between 18-80 years old, suffering from fatigue (as a main symptom) of not yet explained origin, which had lasted for at least 2 weeks, but no longer than 2 years.

Using questionnaires, data on patients, diagnosis, treatment, and outcomes was collected from physicians and patients collected for the differential diagnosis in unexplained fatigue symptoms.

For those physicians randomized to the FDDA group data from the FDDA itself was collected.

Data was collected by the participating GPs and internists using electronic data capture (eCRFs) or paper forms (CRFs) at first consultation (baseline), and at 1, 2, 3 and 6 months after study enrolment.

It was planned to recruit 144 GPs who would each recruit 1 patient in phase 1 and 3 patients in phase 2, i.e., 144 patients in phase 1 and 432 patients in phase 2, resulting in 576 patients in total.

All endpoints were evaluated based on the intention-to-treat population and repeated for the per-protocol study population. The planned sample size (144 PCP and 432 patients) informed the clustered randomized design and assumed a 15% between-arm difference in binary response, as determined by McNemar's test.

ELIGIBILITY:
Inclusion Criteria:

Physicians:

* Established physicians with specialization in general internal medicine (GP).
* Regular consultation of patients with a complaint of a not yet explained fatigue (between 1 every 2 weeks and 5 per week)

Patients:

* 18 to 80 years old
* Male or female
* Fatigue of not yet explained origin
* The reason for encounter had to be fatigue (as a main symptom) of not yet explained origin, which had lasted for at least 2 weeks, but no longer than 2 years before inclusion.
* Subject (or legally acceptable representative) had provided the appropriate written informed consent. Subject had to provide written informed consent before any study-specific procedures were performed.

Exclusion Criteria:

Physicians:

* Works in/or is related to an iron center (a medical center known to be primarily inclined to prescribing intravenous iron supplements in cases of fatigue)
* Known as being experienced in fatigue or CFS (more than five patients per week) Specialized in psychosomatic medicine (in Switzerland: "Fähigkeitsausweis SAPPM / Attestation ASMPP")
* Physicians having a sub-specialty (other than internists working as GPs in a private practice)
* Participation in the feasibility evaluation (excl. for utilization study)

Patients:

* Subject had known pre-existing anemia
* Subject with previous treatment of fatigue by a medical doctor during the last 3 months
* Subject had any pre-known disease, which is responsible for patient's fatigue with a high probability, according to GP's judgement (e.g., CHF, CKD, IBD, RA, MS, Cancer, etc...).
* Subject was known to take any drugs, which could be responsible for inducing fatigue symptoms, according to GP's judgement (e.g., antihistamines, antidepressants, benzodiazepines, hypnotics, anxiolytics, opioid formulations, etc…).
* Subject had a history of drug or alcohol abuse within 2 years prior to the 1st study visit (V1).
* Subject was currently enrolled or had completed any other clinical trial < 30 days prior to 1st study visit (V1).
* Subject had previously participated in the "The Fatigue Differential Diagnosis Aid (FDDA) for General Practitioners: Feasibility study".

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
PGIC 3 months | 3 months
  Patient Global Impression of Change (PGIC) at 3 months. It reflects any change in patient condition.
  It consists of 7 grade scale:
  "very much improved", "greatly improved", "slightly improved", "no change", "slightly worsened", "greatly worsened", "very much worsened". "Very much improved" being the greater improvement state of the patient condition and "Very much worsened" being the worst change in patient condition.

SECONDARY OUTCOMES:
PGIC 6 months | 6 months
  PGIC: Patient Global Impression of Change. "Very much improved" being the greater improvement state of the patient condition and "Very much worsened" being the worst change in patient's condition) at 6 months.
Fatigue reduction 3 or 6 months | 3 or 6 months
  Percentage of patients having experienced a fatigue reduction ≥1 point (NRS), 3 or 6 months after the first visit.
  (NRS: Numeric Rating Scale from 0-10, 0 = no tiredness/exhaustion, 10 = extreme tiredness/exhaustion).
  Response to comments from PRS reviewer:
  We are evaluating whether the FDDA has a positive impact on fatigue reduction. From the statistical perspective, as a secondary endpoint, we were looking at percentage of patients who experienced fatigue improvement by ≥1 point (NRS: Numeric Rating Scale) at 3 or 6 months. Changing this secondary endpoint from "Reduction" to "Change" will represent a different endpoint secondary endpoint.
Time to improvement | 1 to 6 months
  Time expressed by number of days until improvement of fatigue ≥1 point (NRS: Numeric Rating Scale from 0-10, 0 = no tiredness/exhaustion, 10 = extreme tiredness/exhaustion).
Mean fatigue reduction | 1 to 6 months
  Mean number of points of fatigue reduction. (NRS: Numeric Rating Scale from 0-10, 0 = no tiredness/exhaustion, 10 = extreme tiredness/exhaustion)
PGIC improvement 3 and/or 6 months | 3 and/or 6 months
  Percentage of patients with a PGIC (Patient Global Impression of Change). "Very much improved" being the greater improvement state of the patient condition and "Very much worsened" being the worst change in patient condition) indicating response (=any improvement) at 3 months, 6 months and 3 or 6 months.
GP diagnosis confidence | 1 or 3 months
  GP confidence in the established diagnosis. Confidence in the diagnosis expressed by 5 grade scale: "sure", "probable", "possible", "conceivable", "No diagnosis".
CGIC | 1 or 3 months
  Clinical global impression of change (CGIC): 'very much improved' (score=1), 'greatly improved' (score=2), 'slightly improved' (score=3). 'no change' (score=4), 'slightly worsened' (score=5), 'Greatly worsened' (score=6) 'very much worsened' (score=7).
Patient satisfaction | 1 or 3 months
  Patient satisfaction of quality of care (diagnosis and treatment, evaluation scale 5 grades: very dissatisfied, dissatisfied, neutral, satisfied, very satisfied).
Required visits | 1 or 3 months
  Number of required visits for the same condition.
Specialist referrals | 1 to 6 months
  Number of imaging or health services (specialist referrals) required for the diagnosis (MRI, radiograph, etc.).
Final diagnosis | up to 6 months
  Time to final diagnosis
Physician-reported examinations | 1 month and 3 months
  Number of laboratory investigations, imaging, and psychological evaluations at baseline
Type of diagnosis for fatigue | 1 and 3 months
  Type of diagnosis for fatigue at baseline based on the International Classification of Diseases-10 (ICD-10)
Variety of treatments prescribed for fatigue | 1 and 3 months
  No treatment, only iron replacement therapy, iron replacement therapy combined with other treatments, or only other non-iron replacement treatments reported for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Roland von Kändel, Prof. Dr., Principal Investigator — Universitätsspital Zürich, Switzerland; Edouard Battegay, Prof. Dr., Study Chair — Merian Iselin Klinik, Basel, Switzerland
Locations (1):
- QualiPro Schweiz AG, Kriens, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No
It is not planned to share individual participant data with other researchers.

REFERENCES:
- [Derived] von Kanel R, Neuner-Jehle S, Kressig RW, Guessous I, Krayenbuhl PA, Zimmerli L, Angelilo-Scherer A, Keller T, Elzner C, Pauls K, Morin N, Battegay E. Effects of a novel differential diagnosis aid for managing patients with unexplained fatigue in primary care: a prospective randomized, controlled, open and multicenter study in primary care. BMC Prim Care. 2025 May 24;26(1):183. doi: 10.1186/s12875-025-02873-3. PMID 40413405